CLINICAL TRIAL: NCT04330547
Title: Use of Analgesic Treatment to Reduce Signs of Pain in Patients With Disorders of Consciousness: a Double-blind Placebo-controlled Clinical Study.
Brief Title: Use of Analgesic Treatment to Reduce Signs of Pain in Patients With Disorders of Consciousness.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, PhD, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2019-86; 2009-241 (Other: University hospital-faculty committee)
Record Dates: First submitted 2020-03-09; First posted 2020-04-01 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Disorders of Consciousness; Severe Brain Injury; Post-comatose Non-communicative Patients; Vegetative State; Minimally Conscious State
Keywords: Nociception; Pain; Disorder of Consciousness; Nociception coma scale revised
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries; Persistent Vegetative State; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Analgesic administration (Active Comparator): The analgesic treatment will be tailored to the patient's medication and will be based on 3 levels (based on Ventafridda et al., 1985):
  * Level 1 : Non-opioid analgesics
  * Level 2 : Weak opioids analgesics
  * Level 3 : Strong opioids analgesics
  If the patient is already on pain medications, we will add the lowest effective dose of the level above the level of the regular pain medications of the patient. (e.g. if the patient has no analgesic treatment, he will be given a non-opioid analgesic (level 1). If he already has a level 1 treatment, we will go for level 2 medication. If he has level 2 treatment, we will go for level 3. And if the patient is already at level 3, we will increase the dosage by steps (reference: 5mg oxycodone as first choice for level 3 drugs)). Preferably, the medication will be administered by oral intake or gastrostomy feeding tube. If it is not possible, other routes of administration are allowed.
  Interventions: Drug: Analgesic administration
- Placebo administration (Placebo Comparator): Folavit capsules will be used as a placebo
  Interventions: Drug: Placebo administration

INTERVENTIONS:
Drug: Analgesic administration — * Level 1 : Paracétamol 1g/Acetaminophène 1g, Ibuprofène 600mg, Diclofénac 50mg.
  * Level 2: Tramadol 50mg.
  * Level 3: Oxycodone 5mg, Morphine sulfate 10mg.
  * Increase of a prior level 3 medication :
    1. 1/6 of the total dose of daily level 3 medication (e.g. the patient receives 30mg of oxycodone a day. He will be administered a single dose of 5 mg for the study), defined as a breakthrough dose in the management of chronic pain. To standardize the treatment, the dose of the prior level 3 medication will be converted to oxycodone. Several online tools exist to do the conversion between opioids (e.g. mobile app Orthodose ®).
    2. If the oral intake or the gastrostomy use is not possible, the breakthrough dose will be administered by subcutaneous route. The dose will also be 1/6 of the daily dose and will be converted to injectable morphine. Conversion to injectable morphine will be performed with any equivalence tool (such as the mobile app Orthodose ®)
  Arms: Analgesic administration
Drug: Placebo administration — Folavit (folic acid, 0.4 mg)
  Arms: Placebo administration

SUMMARY:
The purpose of this study is to characterize and improve pain and nociception management in patients with disorders of consciousness (DOC). This project is divided into two phases, a first phase to evaluate pain level and a second phase which consist of a clinical trial to evalute pain medication efficacy.

The main aim is to evaluate the use of the Nociception Coma Scale-Revised (NCS-R) and its cut-off score (i.e., 5) as an assessment and management tool to define guidelines for managing pain in patients with DOC. In this double-blind, placebo-controlled clinical study, we will evaluate the use of analgesic treatments in reducing pain in subacute/chronic patients. The project will also allow us to validate the NCS-R cut-off score defined previously.

DETAILED DESCRIPTION:
The study will be performed within one week (i.e, 7 days) and consists of two phases:

* Phase 1 "Patients selection (D0)": Patients will be assessed by the NCS-R during experimental stimulation (rest, tactile, noxious) and mobilizations (physiotherapy). Patients with potential pain will be included in the phase 2.
* Phase 2 "Analgesic administration (D1 and D2)": double-blind placebo-controlled randomized clinical trial on potential responders identified in phase 1. A medical doctor of our team will suggest to the physician in charge to prescribe the dedicated medication. One placebo and one real treatment will be administered on day 1 and 2 by the nurses at least half-hour before the physiotherapy. Randomization between day 1 and 2 will be applied at that time.

For each day of phase 1 and 2, several assessments will be performed: NCS-R, CRS-R and spasticity assessment.

ELIGIBILITY:
Inclusion Criteria:

* Have had an acquired brain injury with a loss of consciousness > 28 days (patients) or have no history of previous brain injury (healthy controls)
* Legally authorized surrogate available to provide informed consent.
* Diagnosis of vegetative/unresponsive (VS/UWS) or minimally conscious state (MCS) or emergence of the minimally conscious state without communication (eMCS; as defined by the CRS-R, see above).
* Medically stable (i.e., no systemic illness or disease).
* Patients with NCS-R score during mobilization above or equal to the previously determined cut-off score or NCS-R scores during mobilization equivalent to NCS-R score obtain during nociceptive stimulation will be included in the second phase of the study (i.e. D1 and D2).

Exclusion Criteria:

* History of developmental, neurologic, or major psychiatric disorder resulting in functional disability.
* Contraindication or unwillingness to discontinuing sedating and centrally-active drugs (benzodiazepine, long-acting sedating drugs) within 48 hours of assessment.
* Upper limb contusions, fractures or flaccid paralysis.
* Uncontrolled epilepsy and already on level 1 drugs

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Nociception Coma Scale-Revised (NCS-R) | through study completion, an average of 2 years
  The NCS-R (Chatelle et al., 2012) is used to assess the perception of acute pain in patients with disorders of consciousness. It is composed of 3 subscales (motor, verbal and facial expressions) respectively scoring from 0 (no response) to 3 (highest response level). Here the NCS-R is administered in 4 different conditions: at rest, during tactile stimulation, during experimental nociceptive stimulation (pressure on the bed of the left and right nail) and during mobilization (physiotherapy).
Coma Recovery Scale-Revised (CRS-R) | through study completion, an average of 2 years
  The CRS-R (Giacino et al., 2004) is the gold standard for the behavioural assessment of the level of consciousness and is widely used in patients with chronic disorders of consciousness. The CRS-R is composed of six subscales that assess the following domains: visual, motor, auditory and oro-motor/verbal functions, as well as communication, and arousal. The score ranges from 0 to 23, in which the lowest score indicates coma and the highest score indicates the emergence from the minimally conscious state. The diagnosis is made according to the presence\absence of particular behavioural responses.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | through study completion, an average of 2 years
  The MAS (Bohannon et al., 1987) is used to assess spasticity (reflex contraction in response to passive stretching). This is a scoring scale from 0 (no increase in muscle tone) to 4 (very strong increase in tone, stiffness), which will depend on the speed of execution of the movement (the faster the limb will be mobilized the more spastic it will be) and which must be performed at least 3 times for each joint.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Laureys, M.D., P.h.D, Study Director — Centre du Cerveau, Coma Science Group (GIGA Consciousness)
Locations (1):
- Centre Hospitalier Universitaire de Liège, Liège, Belgium

REFERENCES:
- [Background] Ventafridda V, Saita L, Ripamonti C, De Conno F. WHO guidelines for the use of analgesics in cancer pain. Int J Tissue React. 1985;7(1):93-6. PMID 2409039
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342
- [Background] Bohannon RW, Larkin PA, Smith MB, Horton MG. Relationship between static muscle strength deficits and spasticity in stroke patients with hemiparesis. Phys Ther. 1987 Jul;67(7):1068-71. doi: 10.1093/ptj/67.7.1068. PMID 3602099
- [Background] Chatelle C, Majerus S, Whyte J, Laureys S, Schnakers C. A sensitive scale to assess nociceptive pain in patients with disorders of consciousness. J Neurol Neurosurg Psychiatry. 2012 Dec;83(12):1233-7. doi: 10.1136/jnnp-2012-302987. Epub 2012 Aug 20. PMID 22906615